CLINICAL TRIAL: NCT04534816
Title: Feasibility and Usability of Intraoperative Fluorescent Angiography With Indocyanine Green in Penetrating Abdominal Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, JENS OSTERKAMP, M.D, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11068
Record Dates: First submitted 2020-08-24; First posted 2020-09-01 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Abdominal Injuries
Keywords: ICG; intestinal injury; gunshot
MeSH Terms: conditions — Abdominal Injuries

STUDY DESIGN:
Intervention Model Description: Pending patient acceptance all are eligible for inclusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Indocyanine Green (Experimental): patients abdominal injuries and repair will be investigated using Indocyanine Green
  Interventions: Diagnostic Test: Indocyanine Green

INTERVENTIONS:
Diagnostic Test: Indocyanine Green — Perfusion assessments

SUMMARY:
The surgical management of penetrating bowel and intestinal injuries, inflicted via a gunshot or knife stabbing, has long been a topic of debate [1-3]. The surgical management principally consists of: (i) primary repair; (ii) primary diversion or (iii) an initial abbreviated so called "damage control" operation followed by a definitive surgical intervention once the patient is stabilized [4-9] . Different classifications systems have been proposed to help determine the best operative option [2,3,10-14], but intestinal injuries can be difficult to manage and despite improvements in the diagnostics and treatment of penetrating abdominal trauma, high mortality and morbidity rates are prevalent [15,16]. In order to determine the correct surgical option an accurate determination of intestinal viability is essential. But clinically assessing regional perfusion is challenging and surgeons' clinical risk assessment of anastomotic leaks have shown a low predictive value [17]. Hence, there is a need for more precise diagnostic tool helping the surgeon in assessing intestinal viability the extent of intestinal injury.

Indocyanine green (ICG) fluorescence angiography (ICG-FA) is an applied method for to assessing visceral perfusion worldwide. The obtained fluorescent signal after intravenous injection, is considered proportional to blood flow, thus aiding the surgeon to detect and address inadequate regional perfusion, despite satisfactory macroscopic appearance, intraoperatively [18-21]. Hence, the use of perioperative ICG-FA, has reduced the risk of anastomotic leaks after esophageal and colorectal surgery [22-25] and in the setting of acute mesenteric ischemia, significantly reduced the extent of intestinal resection [26]. In retrospective review of 186 war related trauma cases the use of ICG-FA was deemed useful however only 9 of these cases were truncal/abdomen/gastrointestinal and no objective definition of usability was provided [27]. Hence, data on the usability and feasibility of ICG-FA for in penetrating abdominal trauma is limited and to our knowledge has not been investigate in a civilian population previously.

The present study aimed to investigate the usability and feasibility of ICG-FA in patients undergoing open abdominal exploration for penetrating abdominal trauma

DETAILED DESCRIPTION:
The surgical management of penetrating bowel and intestinal injuries has been the topic of debate since before the second world war [1-3]. The injury is most often inflicted via a gunshot or knife stabbing. Different classifications systems have been proposed to help determine the best operative option: (i) Flint Grading System (FGS); (ii) Penetrating Abdominal Trauma Index (PATI); (iii) Colonic/Rectal Injury Scale (CIS/RIS); and (iv) destructive/non-destructive colonic injuries; (v) Stone and Fabian's criteria [2,3,10-14].

Principally, a penetrating injury of the intestine can be managed by: (i) primary repair (suturing the hole in the intestine); (ii) primary diversion (the intestine, above the injury, is brought through the abdominal wall as a "stoma") or (iii) an abbreviated primary operation (laparotomy, where large bleeding is stopped and destroyed tissue is removed) and planned reoperation, within 24-48 hours, for definitive treatment (final treatment, for example reconnecting intestinal ends). The concept of abbreviated primary operation, also known as "damage control surgery", is today well established in trauma care [4-6]. A damage control operation with regards to intestinal injury, entails a primary resection/removal of the affected intestinal segment in which the remaining intestinal ends are closed off and not surgically connected (anastomosed) in the first operation.[4-9]. The abdomen is left "open" (the incision through the abdominal wall is not sutured closed but covered with a temporary dressing), and a relaparotomy (re-operation) is conducted once the patient is stabilized (at the end of which the abdominal wall is closed), usually after 24-48 h [4-9]. During the re-laparotomy, the intestines will then either be anastomosed (re-connected), or a stoma will be created if the intestine is deemed too damaged to be re-connected [4-9].

Non-destructive colonic injuries (Flint grades 1 & 2 and CIS grades I to III) are generally treated with primary repair, which involves the identification, debridement and single-layer suture repair of perforation and then dressing the repaired site with omentum (an intra-abdominal layer of fat and vessels) [1,2,10,12]. Primary repair is generally considered the better option in this setting [1-3,28].

Destructive colon wounds (Flint grade 3 or CIS grades IV and V) encompass those injuries that require segmental resection (parts of the large intestine have to be removed) due to extensive damage or loss of blood supply or both [10,12]. The management of destructive colon wounds is less clear and is still debatable. However, primary repair has been deemed as a safe option, while primary diversion has been opted for in particular cases [1-3,9,11,29-33]. In unstable patients; those with hypovolemic shock (large blood loss), blood-poisoning due to intestinal content leaking into the abdominal cavity, systemic hypothermia (low body temperature), and complex intra-abdominal injuries; an abbreviated laparotomy is considered to be an appropriate course of action [7,11,30,32-34].

In colonic trauma, the anastomosis leak rate (the connection between to intestinal ends breaks down) is reported between 4-27% [34-37]. A leak in the sight of intestinal connection is a severe complication which greatly increases the length of hospitalization, increases patient morbidity and has a significant negative impact on patient's recovery. The mortality rate for an anastomotic leak around 10-15% [38,39]. Factors associated with anastomotic failure include co-morbid immune-compromising disorders such as diabetes mellitus, acquired immunodeficiency syndrome, cirrhosis and a transfusion requirement of more than six units of blood [36]. Other potential risk factors appear to be shock, significant associated injuries, and delay of operation [35,36].

In firearm injuries the tissue damage is proportionate to a variety of factors: Projectile velocity, -entrance profile, -calibre, -design, distance travelled within the body (penetrating projectiles deliver their total kinetic energy to the body, whereas perforating projectiles transfer significantly less), biologic characteristics of the impacted tissue and the mechanisms of tissue disruption (e.g. stretching, tearing, crushing) [40]. The extent of damage in the tissue surrounding the entered organ can be difficult to assess, and despite improvements in diagnostics and treatment of abdominal gunshot wounds, high mortality and morbidity rates are still found [15,16].

In conclusion, intestinal injuries can be difficult to manage. A primary repair is preferable but there is a need for more precise diagnostic tools helping the surgeon to access the extent of intestinal injury. Also, reducing the extent of intestinal removal has a high value for the patient as extensive resections can lead to nutritional difficulties even after discharge.

Fluorescence guided surgery Assessing intestinal blood supply is a challenging task even for experienced surgeons. One of the biggest concerns is the blood supply of the anastomosis (the surgical connection between to intestinal ends) since poor blood supply is regarded as a significant risk factor for anastomotic leak [41-44]. As mentioned above, an anastomotic leak is a severe complication in gastrointestinal surgery and has a significant negative impact on patients recovery with the mortality rate for an anastomotic leak around 10-15% [38,39].

Fluorescence guided surgery (FGS) enables visualization of structures that are otherwise hidden from the naked human eye. A fluorescent contrast agent is used, most often indocyanine green (ICG), and by illuminating the tissue with near-infrared light, the excited ICG can be detected by a camera with an optical filter. ICG is a tricarbocyanine dye with very few adverse events, a short half-life, and exclusively metabolized in the liver and excreted unchanged in the bile [45,46]. The safety of ICG well established and the contrast is used routinely in surgical settings worldwide, just as it has gained popularity in oncological surgery in recent years [45-47].

ICG binds to plasma proteins in the blood after intravascular injection, and by illuminating the tissue with near-infrared red light, the fluorescence intensity during the first passage in tissue is considered proportional to blood flow (perfusion). This real-time visualization of visceral perfusion (blood flowing to a given organ) may reduce the rate of anastomotic leakage because inadequate vascularization can be detected during the operation [18-20]. Also, the option for intraoperative visual assessment of blood flow to the intestine, stomach and surrounding tissues, allowing for modification to the surgical plan, may eliminate anastomotic break down or leak due to inadequate vascularization despite satisfactory blood supply on naked-eye appearance [20,21,48], (Figure 1).

Figure 1. A. Intestinal segment as viewed with the naked eye. B. Evaluation of blood flow after injection of ICG, viewed with the infra-red camera (ICG-FA). C. A computer generated combination of images A and B ("overlay") allowing the surgeon to evaluate intestinal blood supply.

In a prospective observational study on patients with a left-sided colorectal cancer, ICG fluorescence angiogram (FA) altered operative decisions in 34.5% of the cases (n=111) i.e. the site of resection was adapted after tissue perfusion evaluated with ICG FA. Also, the use of ICG FA significantly reduced the anastomotic leak rate in patients undergoing surgery for colorectal cancer [49]. In patients undergoing esophagectomy, the use of ICG FA with intervention was found to have a risk reduction for complications of 69% and a significantly lowered risk of anatomic leaks [25].

The use of ICG FA has been shown to improve patient outcome and reduce patients risks in elective settings, however, there is much need for evaluation in the acute/emergency setting. The risk of complications, patient morbidity and mortality are inherently higher in an emergency surgical setting compared to an elective/planned setting [50]. Thus, it is feasible to believe that the use of ICG FA in an emergency setting will improve patient outcome and reduce risk of complications. There is to date little literature on the use of ICG FA in an emergency/trauma setting. However, a recent retrospective study by Karampinis et al. 2018 deemed the use of ICG FA as a feasible and technically reliable technique in patients undergoing emergency surgery for acute mesenteric ischemia. Indocyanine Green FA provided additional information regarding intestinal perfusion in 18 of their 53 cases (35%). In 11 patients the surgical strategy was amended by ICG angiography, showing adequate perfusion, and thus no indication for intestinal resection. No further resections were performed on these patients during the second- and third- look laparotomies [26]. In March 2015, Green et al. presented a retrospective review of all war-related traumatic and reconstructive cases employing the intraoperative use of indocyanine green angiography within the US army over a three year period [27]. They concluded that - Intraoperative fluorescent angiography is an objective, useful tool to assess various war-related traumatic injuries [27].

The Department of Surgical Gastroenterology, Rigshospitalet, Denmark, have developed an ICG quantification algorithm which has been validated and described earlier [51]. This algorithm has now been incorporated into a touch screen tablet, allowing for live perioperative quantitative perfusion assessments with ICG (Q-ICG). A color-coded map of perfusion intensity is provided as an overlay on the white light visualized tissue (Figure 2). In a feasibility study of ten patients undergoing surgery for stomach cancer, significant alterations of optimal perfusion points selected by surgeons were found when comparing points selected in white light, ICG FA and Q-ICG (Nerup, in review).

Figure 2. The remaining stomach (gastric conduit) viewed by white light, Near-Infrared Light (ICG FA) and with Q-ICG overlay.

As ICG FA can assess micro-perfusion, we believe that it has the possibility to improve intraoperative evaluation of tissue integrity and as such improve the surgical plan and outcome in patients suffering gunshots to the abdominal viscera. We also believe that the quantification tool provided by Rigshospitalet will further assist the surgical decision-making.

Aim This study aims to evaluate the feasibility of perfusion assessment with traditional visual, visual ICG FA and Q-ICG.

referenses

1. Cheong JY, Keshava A. Management of colorectal trauma: a review. ANZ J Surg. 2017;87(7-8):547-53.
2. Maxwell RA, Fabian TC. Current management of colon trauma. World J Surg. 2003;27(6):632-9.
3. Greer LT, Gillern SM, Vertrees AE. Evolving colon injury management: a review. Am Surg. 2013;79(2):119-27.
4. Burch JM, Ortiz VB, Richardson RJ, Martin RR, Mattox KL, Jordan GL. Abbreviated laparotomy and planned reoperation for critically injured patients. Ann Surg. 1992;215(5):476-83-4.
5. Hirshberg A, Mattox KL. Planned reoperation for severe trauma. Ann Surg. 1995;222(1):3-8.
6. Hirshberg A, Mattox KL. "Damage control" in trauma surgery. Br J Surg. 1993;80(12):1501-2.
7. Ordoñez CA, Pino LF, Badiel M, Sánchez AI, Loaiza J, Ballestas L, Puyana JC. Safety of performing a delayed anastomosis during damage control laparotomy in patients with destructive colon injuries. J Trauma. 2011;71(6):1512-7-8.
8. Miller PR, Chang MC, Hoth JJ, Holmes JH, Meredith JW. Colonic resection in the setting of damage control laparotomy: is delayed anastomosis safe? Am Surg. 2007;73(6):606-9-10.
9. Tatebe LC, Jennings A, Tatebe K, Handy A, Prajapati P, Smith M, Do T, Ogola GO, Gandhi RR, Duane TM, Luk S, Petrey LB. Traumatic colon injury in damage control laparotomy-A multicenter trial. J Trauma Acute Care Surg. 2017;82(4):742-9.
10. Moore EE, Dunn EL, Moore JB, Thompson JS. Penetrating abdominal trauma index. J Trauma. 1981;21(6):439-45.
11. Sharpe JP, Magnotti LJ, Weinberg JA, Shahan CP, Cullinan DR, Marino KA, Fabian TC, Croce MA. Applicability of an Established Management Algorithm for Destructive Colon Injuries after Abbreviated Laparotomy: A 17-Year Experience. J Am Coll Surg. 2014;218(4):636-41.
12. Flint LM, Vitale GC, Richardson JD, Polk HC. The injured colon: relationships of management to complications. Ann Surg. 1981;193(5):619-23.
13. Stone HH, Fabian TC. Management of perforating colon trauma: randomization between primary closure and exteriorization. Ann Surg. 1979;190(4):430-6.
14. Moore EE, Cogbill TH, Malangoni MA, Jurkovich GJ, Champion HR, Gennarelli TA, McAninch JW, Pachter HL, Shackford SR, Trafton PG. Organ injury scaling, II: Pancreas, duodenum, small bowel, colon, and rectum. J Trauma. 1990;30(11):1427-9.
15. Fackler ML. Civilian gunshot wounds and ballistics: dispelling the myths. Emerg Med Clin North Am. 1998;16(1):17-28.
16. Swan KG, Swan RC. Principles of ballistics applicable to the treatment of gunshot wounds. Surg Clin North Am. 1991;71(2):221-39.
17. Karliczek A, Harlaar NJ, Zeebregts CJ, Wiggers T, Baas PC, van Dam GM. Surgeons lack predictive accuracy for anastomotic leakage in gastrointestinal surgery. Int J Colorectal Dis. 2009;24(5):569-76.
18. Mangano A, Fernandes E, Gheza F, Bustos R, Chen LL, Masrur M, Giulianotti PC. Near-Infrared Indocyanine Green-Enhanced Fluorescence and Evaluation of the Bowel Microperfusion During Robotic Colorectal Surgery: a Retrospective Original Paper. Surg Technol Int. 2019;34.
19. Zehetner J, DeMeester SR, Alicuben ET, Oh DS, Lipham JC, Hagen JA, DeMeester TR. Intraoperative Assessment of Perfusion of the Gastric Graft and Correlation With Anastomotic Leaks After Esophagectomy. Ann Surg. 2015;262(1):74-8.
20. Mangano A, Gheza F, Chen LL, Minerva EM, Giulianotti PC. Indocyanine Green (Icg)-Enhanced Fluorescence for Intraoperative Assessment of Bowel Microperfusion During Laparoscopic and Robotic Colorectal Surgery: The Quest for Evidence-Based Results. Surg Technol Int. 2018;32:101-4.
21. Gossedge G, Vallance A, Jayne D. Diverse applications for near infra-red intraoperative imaging. Color Dis. 2015;17:7-11.
22. Watanabe J, Ishibe A, Suwa Y, Suwa H, Ota M, Kunisaki C, Endo I. Indocyanine green fluorescence imaging to reduce the risk of anastomotic leakage in laparoscopic low anterior resection for rectal cancer: a propensity score-matched cohort study. Surg Endosc. 2019;
23. Sujatha-Bhaskar S, Jafari MD, Stamos MJ. The Role of Fluorescent Angiography in Anastomotic Leaks. Surg Technol Int. 2017;30:83-8.
24. Alekseev M, Rybakov E, Shelygin Y, Chernyshov S, Zarodnyuk I. A Study investigating the Perfusion of Colorectal Anastomoses Using FLuorescence AnGiography: results of FLAG randomized trial. Color Dis. 2020;
25. Ladak F, Dang JT, Switzer N, Mocanu V, Tian C, Birch D, Turner SR, Karmali S. Indocyanine green for the prevention of anastomotic leaks following esophagectomy: a meta-analysis. Surg Endosc. 2019;33(2):384-94.
26. Karampinis I, Keese M, Jakob J, Stasiunaitis V, Gerken A, Attenberger U, Post S, Kienle P, Nowak K. Indocyanine Green Tissue Angiography Can Reduce Extended Bowel Resections in Acute Mesenteric Ischemia.
27. Green JM, Sabino J, Fleming M, Valerio I. Intraoperative Fluorescence Angiography: A Review of Applications and Outcomes in War-Related Trauma. Mil Med. 2015;180(3S):37-43.
28. Choi WJ. Management of colorectal trauma. J Korean Soc Coloproctol. 2011;27(4):166-72.
29. Nelson RL, Singer M. Primary repair for penetrating colon injuries. Cochrane Database Syst Rev. 2003;(3).
30. Bhimji SS, Burns B. Penetrating Abdominal Trauma [Internet]. StatPearls. StatPearls Publishing; 2018.
31. Mansor S, Bendardaf R, Bougrara M, Hagam M. Colon diversion versus primary colonic repair in gunshot abdomen with penetrating colon injury in Libyan revolution conflict 2011 (a single center experience). Int J Colorectal Dis. 2014;29(9):1137-42.
32. Smith IM, Beech ZKM, Lundy JB, Bowley DM. A prospective observational study of abdominal injury management in contemporary military operations: damage control laparotomy is associated with high survivability and low rates of fecal diversion. Ann Surg. 2015;261(4):765-73.
33. Shazi B, Bruce J, Laing G, Sartorius B, Clarke D. The management of colonic trauma in the damage control era. Ann R Coll Surg Engl. 2017;99(1):76-81.
34. Ott MM, Norris PR, Diaz JJ, Collier BR, Jenkins JM, Gunter OL, Morris JA. Colon Anastomosis After Damage Control Laparotomy: Recommendations From 174 Trauma Colectomies. J Trauma Inj Infect Crit Care. 2011;70(3):595-602.
35. Murray JA, Demetriades D, Colson M, Song Z, Velmahos GC, Cornwell EE, Asensio JA, Belzberg H, Berne T V. Colonic resection in trauma: colostomy versus anastomosis. J Trauma. 1999;46(2):250-4.
36. Demetriades D, Murray JA, Chan L, Ordoñez C, Bowley D, Nagy KK, et al. Penetrating colon injuries requiring resection: diversion or primary anastomosis? An AAST prospective multicenter study. J Trauma. 2001;50(5):765-75.
37. Gingold DS, Murrell ZA, Fleshner PR. A Prospective Evaluation of the Ligation of the Intersphincteric Tract Procedure for Complex Anal Fistula in Patients With Crohn's Disease. Ann Surg. 2014;260(6):1057-61.
38. Vallance A, Wexner S, Berho M, Cahill R, Coleman M, Haboubi N, Heald RJ, Kennedy RH, Moran B, Mortensen N, Motson RW, Novell R, O'Connell PR, Ris F, Rockall T, Senapati A, Windsor A, Jayne DG. A collaborative review of the current concepts and challenges of anastomotic leaks in colorectal surgery. Colorectal Dis. 2017;19(1):O1-12.
39. Hyman N, Manchester TL, Osler T, Burns B, Cataldo PA. Anastomotic leaks after intestinal anastomosis: it's later than you think. Ann Surg. 2007;245(2):254-8.
40. Bartlett CS, Helfet DL, Hausman MR, Strauss E. Ballistics and gunshot wounds: effects on musculoskeletal tissues. J Am Acad Orthop Surg. 8(1):21-36.
41. Pommergaard H-C, Achiam MP, Burcharth J, Rosenberg J. Impaired blood supply in the colonic anastomosis in mice compromises healing. Int Surg. 2015;100(1):70-6.
42. Kruschewski M, Rieger H, Pohlen U, Hotz HG, Buhr HJ. Risk factors for clinical anastomotic leakage and postoperative mortality in elective surgery for rectal cancer. Int J Colorectal Dis. 2007;22(8):919-27.
43. Kim MJ, Shin R, Oh H-K, Park JW, Jeong S-Y, Park J-G. The impact of heavy smoking on anastomotic leakage and stricture after low anterior resection in rectal cancer patients. World J Surg. 2011;35(12):2806-10.
44. Fawcett A, Shembekar M, Church JS, Vashisht R, Springall RG, Nott DM. Smoking, hypertension, and colonic anastomotic healing; a combined clinical and histopathological study. Gut. 1996;38(5):714-8.
45. Staller BJ, Staller BJ, Hepner G, Banka VS, Finney RA. Adverse Reactions After Administration of Indocyanine Green. JAMA J Am Med Assoc. 1978;240(7):635.
46. Alander JT, Kaartinen I, Laakso A, Pätilä T, Spillmann T, Tuchin V V., Venermo M, Välisuo P. A Review of Indocyanine Green Fluorescent Imaging in Surgery. Int J Biomed Imaging. 2012;2012:1-26.
47. Baiocchi GL, Diana M, Boni L. Indocyanine green-based fluorescence imaging in visceral and hepatobiliary and pancreatic surgery: State of the art and future directions. World J Gastroenterol. 2018;24(27):2921-30.
48. Boni L, Fingerhut A, Marzorati A, Rausei S, Dionigi G, Cassinotti E. Indocyanine green fluorescence angiography during laparoscopic low anterior resection: results of a case-matched study. Surg Endosc. 2017;31(4):1836-40.
49. Blanco-Colino R, Espin-Basany E. Intraoperative use of ICG fluorescence imaging to reduce the risk of anastomotic leakage in colorectal surgery: a systematic review and meta-analysis. Tech Coloproctol. 2018;22(1):15-23.
50. Mullen MG, Michaels AD, Mehaffey HJ, Guidry CA, Turrentine LE, Hedrick TL, Friel CM. Risk associated with complications and mortality after urgent surgery vs elective and emergency surgery : Implications for defining "quality" and reporting outcomes for urgent surgery. JAMA Surg. 2017;152(8):768-74.
51. Nerup N, Andersen HS, Ambrus R, Strandby RB, Svendsen MBS, Madsen MH, Svendsen LB, Achiam MP. Quantification of fluorescence angiography in a porcine model. Langenbeck's Arch Surg. 2017;402(4):655-62.
52. Owens SL. Indocyanine green angiography. Br J Ophthalmol. 1996;80(3):263-6.
53. Spinoglio G, Bertani E, Borin S, Piccioli A, Petz W. Green indocyanine fluorescence in robotic abdominal surgery. Updates Surg. 2018;70(3):375-9.

ELIGIBILITY:
Inclusion Criteria:

* Patients (above 18 years) scheduled for emergency laparotomy due to penetrating abdominal trauma

Exclusion Criteria:

* Allergy towards; iodine, indocyanine green or shellfish
* Liver insufficiency
* Thyrotoxicosis
* Pregnancy or lactation
* Legally incompetent for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility and usability of ICG-FA | through study completion, an average of 1 year
  Feasibility is defined as the completion rates of the ICG angiography. For each ICG assessment, the operating surgeon will be asked to fill out the widely used System Usability Scale (SUS®).

SECONDARY OUTCOMES:
Surgical management | through study completion, an average of 1 year
  If the use of ICG addes intraoperative information which influences the choice of surgical management, this will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Achiam, DMSci, Study Director — Rigshospitalet, Denmark
Locations (1):
- Tygerberg Hospital, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel MQ, Osterkamp JT, Buitendag JJ, Forgan TR, Steyn E. Indocyanine green fluorescence angiography in the management of intestinal injuries following penetrating abdominal trauma: a case-control study comparing postoperative outcomes. Int J Surg. 2024 Dec 1;110(12):7624-7629. doi: 10.1097/JS9.0000000000002096. PMID 39434689